CLINICAL TRIAL: NCT03429127
Title: Comparison of Normal Saline and Balanced Crystalloid Intravenous Therapy During Neurosurgery
Brief Title: Normal Saline Vrs Balanced i.v. Fluids in Neurosurgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: Sisters of Mercy University Hospital (Other)
Responsible Party: Principal Investigator, Natasa Kovac, Natasa Kovac, M.D., Anesthesiologyst and intensive care medicine subspecialist, Clinical Hospital Centre Zagreb
Other Study IDs: 02/21 AG
Record Dates: First submitted 2018-02-03; First posted 2018-02-12 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Benign Neoplasms; Vascular Malformations, Brain
Keywords: balanced fluids, neurosurgery, plasma osmolality
MeSH Terms: conditions — Neoplasms; Central Nervous System Vascular Malformations | interventions — Saline Solution; Plasma-lyte 148

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal saline fluid group: The patients in this group will receive up to 2000 ml of normal saline during neurosurgical operation.
  Interventions: Other: Normal saline
- Balanced fluid group: The patients in this group will receive up to 2000 ml of balanced fluids during neurosurgical operation.
  Interventions: Other: Balanced fluid

INTERVENTIONS:
Other: Normal saline — Plasma osmolality, acid base status and electrolytes after application up to 2000 ml of normal saline during neurosurgical operation
  Other Names: 0,9 % sodium chloride
  Groups: Normal saline fluid group
Other: Balanced fluid — Plasma osmolality, acid base status and electrolytes after application of up to 2000 ml balanced fluids during neurosurgical operation
  Other Names: Plasma-Lyte 148
  Groups: Balanced fluid group

SUMMARY:
The purpose of this study was to investigate whether the balanced fluids therapy change plasma osmolality in neurosurgical procedures due to brain tumors, meningeomas and arterio-venous malformation.

DETAILED DESCRIPTION:
Normal saline or 0.9% sodium chloride solution is the most commonly used intravenous fluid worldwide and its composition are 154 mmol Na+ and 154 mmol Cl- per litter with osmolality of 308 mOsmol/L. That composition is not "normal" because plasma contains potassium in range between 137-146 mmol/L, and chloride in range between 98-106 mmol/L, with plasma osmolality of 280-295 mOsmol/kg. Recently published data suggested detrimental effects of chloride rich fluids on renal blood flow and glomerular filtration rate, urine output and acute kidney injury. One alternative to saline solution is a buffered, balanced, crystalloid solution with an electrolyte composition similar to plasma and osmolality between 286-295 mOsmol/L. Someone could indicate that such balanced solutions are not suitable for neurosurgical patients because of a possible impact on the brain edema development.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain tumor, meningeomas and vascular malformation.

Exclusion Criteria:

* Patients with signs of elevated intracranial pressure; History of kidney disease, History of heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent neurosurgical procedure because of brain tumor, meningeoma and vascular malformation. And without signs of elevated intracranial pressure and any history of kidney or heart disease.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-10-23 (Estimated); Study Completion 2020-02-23 (Estimated)

PRIMARY OUTCOMES:
Changes in acid base pH status | During operation and immediately after operation
  Changes in acid base pH status after each 500 ml of normal saline vrs. balanced fluid

SECONDARY OUTCOMES:
Changes in electrolytes (sodium and chloride) | During operation and immediately after operation
  Electrolytes changes (sodium and chloride) after each 500 ml of normal saline vrs. balanced fluid

OTHER OUTCOMES:
Plasma osmolality | Immediately after operation
  Whether the applied fluids affect plasma osmolality

CONTACTS AND LOCATIONS:
Overall Officials: Natasa Kovac, M.D., Principal Investigator — UHC Zagreb
Locations (1):
- UHC Zgagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No